CLINICAL TRIAL: NCT06727916
Title: Evaluation of Efficacy and Cost-effectiveness of Brief Behavioral Therapy for Chronic Insomnia Patients Under Medication Treatment At Nguyen Trai Hospital, Ho Chi Minh City
Brief Title: A Randomized, Single-Blind Study Evaluating the Efficacy and Cost-Effectiveness of Brief Behavioral Therapy for Chronic Insomnia Patients Under Medication Treatment At Nguyen Trai Hospital, Ho Chi Minh City
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nguyen Trai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2610/ĐHYD-HĐĐĐ; 2610/ĐHYD-HĐĐĐ (Other: University of Medicine and Pharmacy at Ho Chi Minh City)
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Chronic Insomnia Disorder; Chronic Insomnia; BBT-I; CBT-I
Keywords: Chronic insomnia disorder; chronic insomnia; BBT-I; CBT-I
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BBT-I Group (Experimental): Participants in the intervention group will receive BBT-I in 4 consecutive sessions in addition to standard care.
  Interventions: Behavioral: BBT-I
- Control Group (Other): Patients in the control group will receive standard care.
  Interventions: Other: Non BBT-I

INTERVENTIONS:
Behavioral: BBT-I — Participants in the intervention group will receive BBT-I in 4 consecutive sessions in addition to standard care. Healthcare provider provided BBT-I to the patients.
  Arms: BBT-I Group
Other: Non BBT-I — Patients in the control group will receive standard care.
  Arms: Control Group

SUMMARY:
Insomnia disorder is considered quite common and is recognized as a risk factor for psychiatric disorders. In industrialized countries, chronic insomnia disorder is estimated to affect about 5-10% of the population, with some studies indicating that this rate can reach up to 33% among adults. Research in the Netherlands has shown that insomnia symptoms increase the risk of developing, relapsing, and prolonging mood disorders in men and are associated with recurrent anxiety disorders in women. Without treatment, insomnia disorders are challenging to improve and can impact patients' economic stability and health. Treating insomnia can support recovery and prevent mental disorders, particularly mood disorders.

One of the commonly referenced non-pharmacological treatments for insomnia worldwide is Cognitive Behavioral Therapy for Insomnia (CBT-I). This therapy has been recognized by the American College of Physicians as a first-line and highly effective treatment for insomnia. However, it still faces several barriers to widespread application in clinical practice, such as resource constraints and the time commitment required from patients. As a result, some studies abroad have shown that physicians may be reluctant to recommend CBT-I alone, even though it is considered the preferred treatment. To address these challenges, numerous international studies have expanded the range of providers (such as pharmacists and nurses) or adopted shortened versions, such as Brief Behavioral Treatment for Insomnia (BBT-I), in hospitals or community pharmacies. BBT-I has been proven effective among older adults with a 2+2 design (two in-person sessions and two follow-up calls) and among younger adults using an electronic format. This is a brief, evidence-based therapy designed to encourage the application of CBT-I techniques in primary healthcare settings, demonstrating effectiveness when performed by healthcare providers with basic training. A significant advantage of combining CBT-I and BBT-I in treating insomnia is the reduction in medication use. When effectively implemented, it can shorten treatment duration, reduce hospitalization rates, decrease adverse effects from drug interactions, and improve patients' quality of life, ultimately reducing the financial burden on healthcare facilities and improving the quality of medical services.

In Vietnam, CBT-I and BBT-I therapies are not yet widely applied or popularized. Based on the current situation and the desire to apply these therapies in treating chronic insomnia patients to improve quality of life and reduce medication costs, in 2023, Nguyen Trai Hospital collaborated with Thong Nhat Hospital and the Saigon Center for Pharmaceutical Science and Technology to conduct a city-level scientific and technological research program on the application of BBT-I in supporting the treatment of chronic insomnia in the elderly. The research developed a "Sleep Support Guide" as a resource for healthcare workers to counsel patients and provide essential information related to insomnia. Results from the study also showed that BBT-I could help improve sleep-related parameters, life quality, and sleep quality among elderly patients. However, the study had some limitations, such as being conducted only on elderly subjects, with a follow-up period of one month post-intervention for sleep parameters and three months for medication usage metrics, without a cost-effectiveness comparison with medication-only treatments. Therefore, further in-depth research with a wider range of subjects and a comparison with standard hospital treatments is necessary for broader application of this method in practice.

Objective 1: To investigate the characteristics of chronic insomnia patients receiving medication at Nguyen Trai Hospital in Ho Chi Minh City.

Objective 2: To assess the effectiveness of BBT-I in improving sleep quality and quality of life after one and three months compared to non-application in chronic insomnia patients receiving medication at Nguyen Trai Hospital in Ho Chi Minh City.

Objective 3: To evaluate the cost-effectiveness of BBT-I in improving sleep quality and quality of life when applied to chronic insomnia patients receiving medication at Nguyen Trai Hospital in Ho Chi Minh City.

ELIGIBILITY:
Inclusion Criteria:

The study includes patients who fully meet the following criteria:

Patients with an outpatient prescription diagnosed with "sleep disorder" (ICD-10: G47), insomnia disorder [difficulty initiating and maintaining sleep] (ICD-10: G47.0), nonorganic insomnia (ICD-10: F51.0), or agrypnia [sleep disorder] (ICD-10: U55.621). Diagnoses are based on DSM-5 criteria.

Patients aged 18 years or older. Agreement to participate in the study.

Exclusion Criteria:

Cognitive impairment (inability to understand counseling content). Presence of a triggering factor during the study period (hospitalization, acute exacerbation of comorbid conditions, or a psychological trauma) as these conditions may induce insomnia.

Conditions incompatible with sleep restriction therapy:

Epilepsy. Untreated obstructive sleep apnea (diagnosed or high-risk based on STOP-BANG screening).

Untreated bipolar disorder. Suicidal intent. Parasomnias related to NREM sleep (sleepwalking, night terrors). Diagnosed with other sleep disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in PSQI score | 1 and 3 months
  The PSQI (developed by Buysse) is a standardized tool used to assess both sleep quantity and quality. It includes 19 items that provide a subjective evaluation of sleep metrics such as total sleep time, perceived restfulness, and sleep disturbances.